CLINICAL TRIAL: NCT01120483
Title: Prevalence and Impact of Malnutrition in Hospitalised Patients
Brief Title: Prevalence of Malnutrition in Oncologic Patients
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Kristina Norman, Charite University, Berlin, Germany
Other Study IDs: Onco400
Record Dates: First submitted 2010-05-06; First posted 2010-05-11 (Estimated); Last update posted 2010-05-11 (Estimated); Status verified 2006-10

CONDITIONS: Cancer; Malnutrition
Keywords: mortality; functional status
MeSH Terms: conditions — Neoplasms; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Malnutrition is a common phenomenon in cancer patients. Deteriorated nutritional status is associated with poor clinical outcome. The purpose of this study is to determine the prevalence of hospital malnutrition and its impact on functionality, quality of life and mortality in cancer patients and to test the reference percentiles of phase angle values (Bosy Westphal et al JPEN 2006) as indicator of cancer cachexia and predictor of mortality.

Hypothesis:

The fifth reference percentile of the phase angle norm values is a prognostically relevant cut off value indicating cancer cachexia in terms of malnutrition, fatigue and impaired functional status, as well as predictive of 6-month mortality

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from cancer.
* Patients who have signed a written Informed Consent.

Exclusion Criteria:

* Patients with implanted pacemaker or defibrillator
* Patients with neuromuscular disease or hemiplegia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected in primary care clinics.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2006-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of malnutrition | 1 day
  Phase angle (bioelectrical impedance analysis) Nutritional status(SGA), muscle function (grip strength)

SECONDARY OUTCOMES:
Quality of life | 1 day
  Quality of life is determined with the questionnaire QLQ C-30 of the European Organisation for Research and Treatment of Cancer (EORTC)
Mortality | 6 months
  Patients are going to be contacted via telephone six months after the first assessment. Deceased patients will be determined by the local death register
Depression | 1 day
  Risk for depression is assessed using the Center for Epidemiological Studies Depression Scale (CES-D)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Pirlich, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Gastroenterology, Charité Universitätsmedizin Berlin, Campus Mitte, Berlin, State of Berlin, Germany